CLINICAL TRIAL: NCT03141281
Title: Intervention Comparative Effectiveness for Adult Cognitive Training
Acronym: ICE-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Neil Charness, Principal Investigator, Professor of Psychology, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017.20622
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Aging
Keywords: aging; cognitive ability; IADL; driving; financial fraud; perception; attention; memory

STUDY DESIGN:
Intervention Model Description: Random assignment to one of four treatment groups at study entry
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to study condition when administering the tests to participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BrainHQ (Experimental): Participants will be provided with a laptop computer and enrolled in a commercial web-based cognitive training program, BrainHQ, trained on how to access it, and instructed to complete a fixed number of sessions in 20 hours.
  Interventions: Behavioral: BrainHQ
- Rise of Nations (Experimental): Participants will be provided with a laptop computer with the Rise of Nations video game, be trained in game play, and instructed to play the game for 20 hours
  Interventions: Behavioral: Rise of Nations
- IADL training (Experimental): Participants will be enrolled in American Association of Retired Persons' web-based driver training course, trained on how to access it, and asked to complete the course, estimated to take approximately 6-8 hours. They will also be provided with web-based access to a finance and fraud avoidance training tutorial, instructed on how to access it, and be asked to complete the course, estimated to take approximately 5-7 hours. The two courses combined are estimated to take about 15 hours.
  Interventions: Behavioral: IADL Training
- Active Control (Active Comparator): Participants will be provided with a laptop computer and asked to complete 20 hr of training with Sudoku, crossword puzzles, and word search
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: BrainHQ — BrainHQ
  Arms: BrainHQ
Behavioral: Rise of Nations — Rise of Nations
  Arms: Rise of Nations
Behavioral: IADL Training — IADL Training
  Arms: IADL training
Behavioral: Active Control — Puzzle solving
  Arms: Active Control

SUMMARY:
The study will compare the effect of broad and directed (narrow) technology-based training on basic perceptual and cognitive abilities in older adults and on the performance of simulated tasks of daily living including driving and fraud avoidance.

DETAILED DESCRIPTION:
Participants will be randomly assigned to four training conditions: broad training using either 1) Posit Science's web-based "BrainHQ" or 2) the video game Rise of Nations, or to directed training for 3) Instrumental Activities of Daily Living (IADL) training on both driving, American Association of Retired Persons (AARP)'s web-based older driver training program, and training for fraud avoidance, a web-based tutorial on finance and fraud, or 4) to an active control condition of puzzle solving. Training will take approximately 15-20 hr for each treatment condition. Before training begins, participants will take baseline ability tests of perception, attention, memory, and cognition, activities of daily living, as well as a driving simulator test for hazard perception, and a financial fraud recognition test. They will be tested again on these measures following training completion, and at a one-year follow-up from training completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and above
* Plans to stay in the Tallahassee, Leon County area for the next year
* Valid driver's license and drives at least once a month
* Adequate cognitive ability assessed via telephone interview using the Wechsler Memory Scale III with story A score >6 or story B score >4.

Exclusion Criteria:

* Terminal illness with life expectancy less than 12 months
* Reports or exhibits a disabling visual condition assessed as the inability to read printed material
* Reports or exhibits a disabling speech hearing and comprehension condition assessed by inability to hear and comprehend the screener's instructions
* Reports or exhibits a disabling speech production condition assessed as the inability to respond with comprehensible English speech to the screener's queries
* Reports or exhibits a disabling psychomotor condition assessed as the inability to use a keyboard and pointing device
* Has completed the AARP driver training course
* Has played the Rise of Nations video game
* Has trained with Posit Science's "BrainHQ"
* Has trained on the Mind Frontiers video game.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Charness, PhD, Principal Investigator — Florida State University; Walter Boot, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gray N, Yoon JS, Charness N, Boot WR, Roque NA, Andringa R, Harrell ER, Lewis KG, Vitale T. Relative effectiveness of general versus specific cognitive training for aging adults. Psychol Aging. 2022 Mar;37(2):210-221. doi: 10.1037/pag0000663. Epub 2021 Dec 30. PMID 34968102
- [Derived] Yoon JS, Roque NA, Andringa R, Harrell ER, Lewis KG, Vitale T, Charness N, Boot WR. Intervention Comparative Effectiveness for Adult Cognitive Training (ICE-ACT) Trial: Rationale, design, and baseline characteristics. Contemp Clin Trials. 2019 Mar;78:76-87. doi: 10.1016/j.cct.2019.01.014. Epub 2019 Jan 31. PMID 30711665
- Available data/document: Statistical Analysis Plan: https://osf.io/dp8n5/ — https://osf.io/kq8yz/register/565fb3678c5e4a66b5582f67 — Open Science Foundation registration of Data Analysis Plan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants were consented and completed some baseline measures, but removed themselves from the study before they were randomly assigned to a certain condition. Thus, 238 participants agreed to participate in the study, but only 230 participants appear at baseline across conditions.
Groups:
- IADL Training: Training in instrumental activities of daily living. Participants will be enrolled in American Association of Retired Persons' web-based driver training course, trained on how to access it, and asked to complete the course, estimated to take approximately 6-8 hours. They will also be provided with web-based access to a finance and fraud avoidance training tutorial, instructed on how to access it, and be asked to complete the course, estimated to take approximately 5-7 hours. The two courses combined are estimated to take about 15 hours.
  IADL Training: IADL Training
Period: Overall Study
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Started | 57 | 59 | 56 | 58
Post-Test | 50 | 47 | 50 | 56
Completed | 45 | 38 | 42 | 47
Not Completed | 12 | 21 | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- IADL Training: Participants will be enrolled in AARP's web-based driver training course, trained on how to access it, and asked to complete the course, estimated to take approximately 6-8 hours. They will also be provided with web-based access to a finance and fraud avoidance training tutorial, instructed on how to access it, and be asked to complete the course, estimated to take approximately 5-7 hours. The two courses combined are estimated to take about 15 hours.
  IADL Training: IADL Training
- Total: Total of all reporting groups
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control | Total
Number analyzed (Participants) | 57 | 59 | 56 | 58 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (5.9) | 71.4 (5.7) | 72.4 (5.5) | 70.2 (3.8) | 71.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 36 | 31 | 133
  Male | 24 | 26 | 20 | 27 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 5 | 4 | 7 | 10 | 26
  White | 40 | 41 | 40 | 44 | 165
  More than one race | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 9 | 13 | 8 | 2 | 32
Region of Enrollment [Number; unit: participants]
  United States | 57 | 59 | 56 | 58 | 230

OUTCOME MEASURES:

1. Primary Outcome: Fraud Detection Post Training
Description: Percent confidence that a given vignette describing fraud is actually an example of fraud, measured at baseline and immediately after 4 weeks of training. Participants were given a vignette describing fraud (which was mixed in with vignettes not describing fraud) and were asked to give their percent confidence that this is actually an example of fraud. Higher confidence indicates higher accuracy when detecting fraud, with a minimum of 0 and a maximum of 100. Measures accuracy in discriminating fraud from non-fraud text-based scenarios (using 3 parallel forms).
Time Frame: Baseline, Immediately after 4-week intervention training
Population: Participants were instructed that they could refuse any individual measure, which may influence the participant counts for some measures.
Measure: Mean (Standard Deviation); unit: % confidence fraudulent item is fraud
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
% confidence fraudulent item is fraud
  Baseline | 90.42 (9.03) | 85.84 (18.33) | 84.88 (12.31) | 84.32 (16.95)
  Post Training | 85.91 (13.76) | 86.34 (10.91) | 85.88 (19.37) | 83.84 (14.86)

2. Primary Outcome: Driving Simulator Hazard Perception Post Training
Description: Driving simulator (scenarios including hazards) measures of speed, maximum brake compression, and lane position, at baseline and immediately after 4 weeks of training. These measures provide an estimate of accuracy in driving scenarios that involve hazards in the DriveSafety simulator (using 3 parallel forms). All measures were transformed into Z scores and averaged in order to create a measure of overall driving performance, where higher scores represent more dangerous (worse) driving performance.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: Participants were instructed that they could refuse any individual measure, which may influence the participant counts for some measures. This was particularly pronounced for driving simulator measures because of discomfort and simulator sickness.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 31 | 25 | 28 | 36
z-score
  Composite Driving Baseline | -0.06 (0.41) | 0.26 (0.32) | 0.02 (0.32) | 0.12 (0.38)
  Composite Driving Post Training | 0.09 (0.43) | -0.10 (1.20) | -0.21 (1.13) | 0.11 (0.62)

3. Primary Outcome: Self-reported Difficulty With Instrumental Activities of Daily Living (IADLs) Post Training
Description: Self-reported difficulties in completing instrumental activities of daily living, measured at baseline and immediately after 4 weeks of training, with a minimum score of 0 (indicating no difficulty) and a maximum of 3 (indicating severe difficulty). This is a modified short-form version of the Lawton IADL Items, used in the Multicenter AIDS Cohort Study (MACS).
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
units on a scale
  Baseline | 0.31 (0.87) | 0.26 (0.94) | 0.38 (1.52) | 0.39 (0.95)
  Post Training | 0.35 (1.03) | 0.23 (0.89) | 0.22 (1.42) | 0.21 (0.73)

4. Primary Outcome: Speed of Processing Post Training
Description: Scores from Useful Field of View (UFOV) test and Digit Symbol Substitution Test, at baseline and immediately after 4 weeks of training, which each provide a measure of speed of processing. Raw scores were transformed into z scores, UFOV reaction time scores were inverted, then both UFOV and digit symbol scores were averaged in order to create an estimate of overall speed of processing, where higher scores represent better performance.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 45 | 49 | 56
z-score
  Speed of Processing Baseline | 0.09 (0.87) | 0.03 (0.81) | -0.03 (0.65) | 0.01 (0.79)
  Speed of Processing Post Training | 0.34 (0.85) | 0.16 (0.80) | 0.15 (0.71) | 0.13 (0.87)

5. Primary Outcome: Knowledge About Driving Post Training
Description: Test questions based on the American Association of Retired Persons driving course, measured immediately after 4 weeks of training, with a minimum score of 0 and a maximum score of 3. Higher scores indicate more accurate knowledge of driving related information.
Time Frame: Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
score on a scale | 1.49 (0.74) | 1.53 (0.75) | 2.28 (0.90) | 1.36 (0.77)

6. Primary Outcome: Knowledge About Finances and Fraud Post Training
Description: Test questions based on the Finance and Fraud training tutorial, measured immediately after 4 weeks of training, with a minimum score of 0 and a maximum score of 3. Higher scores indicate more accurate knowledge of finance and fraud related information.
Time Frame: Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
score on a scale | 1.65 (1.01) | 1.62 (1.01) | 2.24 (0.77) | 1.54 (0.95)

7. Primary Outcome: Fraud Detection at One Year
Description: Percent confidence that a given vignette describing fraud is actually an example of fraud, measured at baseline and one year after 4 weeks of training. Participants were given a vignette describing fraud (which was mixed in with vignettes not describing fraud) and were asked to give their percent confidence that this is actually an example of fraud. Higher confidence indicates higher accuracy when detecting fraud, with a minimum of 0 and a maximum of 100. Measures accuracy in discriminating fraud from non-fraud text-based scenarios (using 3 parallel forms).
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % confidence fraudulent item is fraud
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 41 | 47
% confidence fraudulent item is fraud
  Baseline | 90.88 (8.86) | 87.78 (16.38) | 86.30 (11.17) | 84.86 (17.58)
  Follow-up | 87.79 (8.95) | 87.17 (12.87) | 91.84 (7.62) | 85.55 (11.56)

8. Primary Outcome: Driving Simulator Hazard Perception at One Year
Description: Driving simulator (scenarios including hazards) measures of speed, maximum brake compression, and lane position, at baseline and one year after 4 weeks of training. These measures provide an estimate of accuracy in driving scenarios that involve hazards in the DriveSafety simulator (using 3 parallel forms). All measures were transformed into Z scores and averaged in order to create a measure of overall driving performance, where higher scores represent more dangerous (worse) driving performance.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 32 | 22 | 21 | 27
z-score
  Composite Driving Baseline | 0.02 (0.44) | 0.31 (0.25) | -0.06 (0.28) | 0.07 (0.38)
  Composite Driving Follow-up | 0.11 (0.50) | 0.34 (0.32) | 0.19 (0.33) | 0.18 (0.37)

9. Primary Outcome: Self-reported Difficulty With Instrumental Activities of Daily Living (IADLs) at One Year
Description: Self-reported difficulties in completing instrumental activities of daily living, measured at baseline and one year after 4 weeks of training, with a minimum score of 0 (indicating no difficulty) and a maximum of 3 (indicating severe difficulty).This is a modified short-form version of the Lawton IADL Items, used in the Multicenter AIDS Cohort Study (MACS).
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 41 | 47
units on a scale
  Baseline | 0.27 (0.81) | 0.16 (0.44) | 0.10 (0.44) | 0.36 (0.92)
  Follow-up | 0.38 (1.54) | 0.22 (0.63) | 0.10 (0.37) | 0.34 (1.31)

10. Primary Outcome: Speed of Processing at One Year
Description: Scores from Useful Field of View (UFOV) test and Digit Symbol Substitution Test, at baseline and one year after 4 weeks of training, which each provide a measure of speed of processing. Raw scores were transformed into z scores, UFOV reaction time scores were inverted, then UFOV and digit symbol scores were averaged in order to create an estimate of overall speed of processing, where higher scores represent better performance.
Time Frame: Baseline, One-year after 4-week intervention training
Population: Participants were instructed that they could refuse any individual measure, which may influence the participant counts for some measures. Some participants may also have dropped from the study mid-session during testing, which means they may be counted as a drop out in other analyses.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 43 | 48
z-score
  Speed of Processing Baseline | 0.10 (0.89) | 0.12 (0.82) | 0.07 (0.47) | 0.01 (0.81)
  Speed of Processing Follow-up | 0.22 (0.89) | 0.36 (0.57) | 0.15 (0.67) | 0.19 (0.74)

11. Primary Outcome: Knowledge About Driving at One Year
Description: Test questions based on the American Association of Retired Persons driving course, measured one year after 4 weeks of training, with a minimum score of 0 and a maximum score of 3. Higher scores indicate more accurate knowledge of driving related information.
Time Frame: One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 41 | 47
score on a scale | 1.36 (0.83) | 1.46 (0.77) | 1.59 (0.84) | 1.62 (0.74)

12. Primary Outcome: Knowledge About Finances and Fraud at One Year
Description: Test questions based on the Finance and Fraud training tutorial, measured immediately after one year of training, with a minimum score of 0 and a maximum score of 3. Higher scores indicate more accurate knowledge of finance and fraud related information.
Time Frame: One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 41 | 47
score on a scale | 1.53 (0.89) | 1.95 (0.88) | 1.78 (0.88) | 1.55 (0.95)

13. Primary Outcome: Driving Simulator Average Speed Post Training
Description: Average speed in a driving simulator measured at baseline and immediately after 4 weeks of training. Speed is a continuous measure in miles per hour, with a minimum of 0 and no maximum. Speed may indicate risky driving behavior.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Miles Per Hour
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 31 | 25 | 28 | 36
Miles Per Hour
  Speed Baseline | 12.46 (1.87) | 13.46 (1.38) | 12.71 (1.63) | 13.12 (1.47)
  Speed Post Training | 13.25 (1.75) | 12.88 (4.01) | 11.88 (3.90) | 13.21 (2.46)

14. Primary Outcome: Driving Simulator Max Brake Compression Post Training
Description: Maximum brake compression in a driving simulator measured at baseline and immediately after 4 weeks of training. Maximum brake compression measures the most that the brake pedal was compressed during driving, with a minimum of 0 and a maximum of 1. Maximum brake compression may indicate urgent stopping.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 31 | 25 | 28 | 36
units on a scale
  Max Brake Baseline | 0.98 (0.05) | 1.00 (0.00) | 0.99 (0.05) | 1.00 (0.00)
  Max Brake Post Training | 0.99 (0.04) | 0.91 (0.28) | 0.90 (0.27) | 0.97 (0.17)

15. Primary Outcome: Driving Simulator Average Lane Position Post Training
Description: Average lane position in a driving simulator measured at baseline and immediately after 4 weeks of training. Lane position measures the average deviation from the center of a lane while driving (values from -1 to 1), averaged across participants, where 0 represents perfect center, negative scores represent deviation to the left (from 0 to -1), and positive scores represent deviation to the right (from 0 to 1). Lane position indicates vehicle control and safety.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 31 | 25 | 28 | 36
units on a scale
  Lane Position Baseline | -0.43 (0.13) | -0.35 (0.11) | -0.41 (0.12) | -0.40 (0.13)
  Lane Position Post Training | -0.41 (0.16) | -0.39 (0.13) | -0.39 (0.17) | -0.37 (0.12)

16. Primary Outcome: Driving Simulator Average Speed at One Year
Description: Average speed in a driving simulator measured at baseline and one year after 4 weeks of training. Speed is a continuous measure in miles per hour, with a minimum of 0 and no maximum. Speed may indicate risky driving behavior.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Miles Per Hour
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 32 | 22 | 21 | 27
Miles Per Hour
  Speed Baseline | 12.71 (1.89) | 13.76 (1.08) | 13.04 (1.65) | 12.96 (1.40)
  Speed Follow-up | 13.36 (1.54) | 14.08 (0.97) | 13.28 (1.15) | 13.70 (1.46)

17. Primary Outcome: Driving Simulator Max Brake Compression at One Year
Description: Maximum brake compression in a driving simulator measured at baseline and one year after 4 weeks of training. Maximum brake compression measures the most that the brake pedal was compressed during driving, with a minimum of 0 and a maximum of 1. Maximum brake compression may indicate urgent stopping.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 32 | 22 | 21 | 27
units on a scale
  Max Brake Baseline | 0.99 (0.04) | 1.00 (0.00) | 0.99 (0.06) | 1.00 (0.00)
  Max Brake Follow-up | 0.98 (0.06) | 1.00 (0.00) | 1.00 (0.00) | 0.99 (0.04)

18. Primary Outcome: Driving Simulator Average Lane Position at One Year
Description: Average lane position in a driving simulator measured at baseline and one year after 4 weeks of training. Lane position measures the average deviation from the center of a lane while driving (values from -1 to 1), averaged across participants, where 0 represents perfect center, negative scores represent deviation to the left (from 0 to -1), and positive scores represent deviation to the right (from 0 to 1). Lane position indicates vehicle control and safety.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 32 | 22 | 21 | 27
units on a scale
  Lane Position Baseline | -0.41 (0.14) | -0.35 (0.11) | -0.46 (0.09) | -0.41 (0.13)
  Lane Position Follow-up | -0.40 (0.19) | -0.35 (0.14) | -0.37 (0.14) | -0.39 (0.11)

19. Primary Outcome: Useful Field of View Post Training
Description: Useful field of view (UFOV) measured at baseline and immediately after 4 weeks of training. UFOV is measured as a response time in milliseconds, with lower times indicating quicker responses.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 46 | 49 | 56
Milliseconds
  UFOV Baseline | 225.84 (201.81) | 229.08 (242.48) | 228.55 (134.75) | 212.14 (145.31)
  UFOV Post Training | 170.04 (194.38) | 217.47 (192.39) | 210.87 (154.27) | 219.92 (215.25)

20. Primary Outcome: Digit Symbol Substitution Test Post Training
Description: The Digit Symbol Substitution Test measured at baseline and immediately after 4 weeks of training. The Digit Symbol Substitution Test is measured through the number of items completed during a 90 second period, where higher scores indicate faster/better performance.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items completed
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
items completed
  Digit Symbol Baseline | 46.45 (12.49) | 45.36 (10.77) | 44.04 (10.11) | 43.71 (13.22)
  Digit Symbol Post Training | 48.90 (11.87) | 48.66 (10.43) | 46.80 (12.24) | 47.07 (12.79)

21. Primary Outcome: Useful Field of View at One Year
Description: Useful field of view (UFOV) measured at baseline and one year after 4 weeks of training. UFOV is measured as a response time in milliseconds, with lower times indicating quicker responses.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 43 | 48
Milliseconds
  UFOV Baseline | 229.38 (205.25) | 199.58 (229.19) | 206.54 (113.42) | 211.90 (154.92)
  UFOV Follow-up | 200.85 (215.83) | 158.65 (68.70) | 214.71 (152.89) | 192.18 (148.15)

22. Primary Outcome: Digit Symbol Substitution Test at One Year
Description: The Digit Symbol Substitution Test measured at baseline and one year after 4 weeks of training. The Digit Symbol Substitution Test is measured through the number of items completed during a 90 second period, where higher scores indicate faster/better performance.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items completed
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 43 | 48
items completed
  Digit Symbol Baseline | 47.02 (12.76) | 45.65 (10.79) | 44.84 (7.84) | 43.58 (12.74)
  Digit Symbol Follow-up | 48.36 (13.22) | 47.65 (14.97) | 48.05 (9.77) | 46.90 (12.25)

23. Secondary Outcome: Technology Proficiency Post Training
Description: Standardized Z-scores of Computer Proficiency Questionnaire and the Mobile Device Proficiency Questionnaire, at baseline and immediately after 4 weeks of training, which provide measures of technology proficiency. Scores are measured as a self-assessed proficiency, where higher scores indicate a higher proficiency and greater ease using a device on various tasks. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
z-score
  CPQ Baseline | 0.16 (0.95) | 0.21 (0.83) | -0.03 (1.03) | -0.13 (1.14)
  CPQ Post Training | 0.24 (0.90) | 0.16 (0.95) | 0.08 (1.01) | -0.06 (1.20)
  MDPQ Baseline | 0.11 (1.02) | 0.21 (0.90) | -0.07 (1.03) | 0.05 (1.03)
  MDPQ Post Training | 0.23 (1.00) | 0.09 (0.93) | -0.04 (1.07) | 0.07 (1.04)

24. Secondary Outcome: Technology Proficiency at One Year
Description: Standardized Z-scores of Computer Proficiency Questionnaire and the Mobile Device Proficiency Questionnaire, at baseline and one year after 4 weeks of training, which provide measures of technology proficiency. Scores are measured as a self-assessed proficiency, where higher scores indicate a higher proficiency and greater ease using a device on various tasks. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 41 | 47
z-score
  CPQ Baseline | 0.11 (0.97) | 0.35 (0.66) | 0.06 (0.91) | -0.21 (1.20)
  CPQ Follow-up | 0.20 (0.89) | 0.50 (0.70) | 0.29 (0.82) | 0.11 (1.13)
  MDPQ Baseline | 0.03 (1.02) | 0.40 (0.72) | -0.04 (0.95) | -0.01 (1.05)
  MDPQ Follow-up | 0.15 (1.02) | 0.39 (0.86) | 0.20 (1.02) | 0.20 (1.07)

25. Secondary Outcome: Numeracy Post Training
Description: Score on the Berlin Numeracy Test taken at baseline and immediately after 4 weeks of training. Scores represent the number of correct items, where higher scores represent better performance, with a minimum score of 0 and a maximum score of 3.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
score on a scale
  Baseline | 2.41 (1.55) | 2.49 (1.32) | 2.38 (1.50) | 2.39 (1.57)
  Follow-up | 2.45 (1.47) | 2.66 (1.70) | 2.16 (1.65) | 2.48 (1.78)

26. Secondary Outcome: Numeracy at One Year
Description: Score on the Berlin Numeracy Test taken at baseline and one year after 4 weeks of training. Scores represent the number of correct items, where higher scores represent better performance, with a minimum score of 0 and a maximum score of 3.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 43 | 48
score on a scale
  Baseline | 2.36 (1.48) | 2.65 (1.27) | 2.47 (1.52) | 2.52 (1.60)
  Follow-up | 2.40 (1.45) | 2.76 (1.40) | 2.14 (1.81) | 2.52 (1.69)

27. Secondary Outcome: Reasoning Ability Post Training
Description: Standardized Z-scores from Raven's Advanced Progressive Matrices and Letter Sets tests, at baseline and immediately after 4 weeks of training, which provide measures of reasoning ability. Scores represent the number of correct items, where higher scores represent better performance. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 47 | 45 | 49 | 54
z-score
  Raven's Baseline | 0.10 (0.98) | 0.14 (0.94) | -0.18 (0.87) | -0.02 (1.08)
  Raven's Post Training | 0.08 (1.03) | 0.13 (0.97) | -0.01 (1.03) | -0.07 (1.19)
  Letter Sets Baseline | 0.19 (0.88) | -0.07 (0.99) | 0.01 (1.01) | 0.00 (1.06)
  Letter Sets Post Training | 0.24 (0.96) | 0.40 (0.84) | 0.23 (0.97) | 0.21 (1.05)

28. Secondary Outcome: Reasoning Ability at One Year
Description: Standardized Z-scores from Raven's Advanced Progressive Matrices and Letter Sets tests, at baseline and one year after 4 weeks of training, which provide measures of reasoning ability. Scores represent the number of correct items, where higher scores represent better performance. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 43 | 35 | 41 | 45
z-score
  Raven's Baseline | 0.10 (0.94) | 0.14 (0.98) | -0.10 (0.86) | 0.05 (1.05)
  Raven's Follow-up | -0.04 (1.07) | 0.08 (0.91) | 0.01 (1.10) | -0.07 (1.09)
  Letter Sets Baseline | 0.25 (0.85) | -0.07 (0.98) | 0.06 (0.87) | 0.02 (1.10)
  Letter Sets Follow-up | 0.21 (0.99) | 0.36 (0.94) | 0.22 (0.90) | 0.06 (1.14)

29. Secondary Outcome: Memory Ability Post Training
Description: Standardized Z-scores from Hopkins Verbal Learning and Rey Auditory Verbal Learning Tests, at baseline and immediately after 4 weeks of training, which provide measures of memory ability. Scores represent the number of correctly recalled items, where higher scores represent better memory. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
z-score
  Hopkins Baseline | -0.01 (0.89) | 0.04 (0.99) | 0.04 (1.12) | 0.15 (0.88)
  Hopkins Post Training | 0.23 (0.97) | 0.05 (0.95) | -0.12 (1.22) | 0.22 (0.93)
  Rey Baseline | -0.22 (0.94) | 0.04 (1.05) | 0.03 (1.03) | 0.17 (0.96)
  Rey Post Training | -0.03 (1.04) | -0.03 (1.00) | -0.04 (1.10) | 0.24 (1.07)

30. Secondary Outcome: Memory Ability at One Year
Description: Standardized Z-scores from Hopkins Verbal Learning and Rey Auditory Verbal Learning Tests, at baseline and one year after 4 weeks of training, which provide measures of memory ability. Scores represent the number of correctly recalled items, where higher scores represent better memory. Scores are standardized using z-scores, with the average at the baseline representing 0, and 1 representing one standard deviation above the average baseline score.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 43 | 48
z-score
  Hopkins Baseline | 0.06 (0.88) | 0.10 (0.86) | 0.16 (0.98) | 0.25 (0.86)
  Hopkins Follow-up | 0.19 (1.00) | 0.21 (0.79) | 0.21 (1.15) | 0.40 (0.87)
  Rey Baseline | -0.18 (0.96) | 0.06 (1.01) | 0.16 (1.02) | 0.21 (0.97)
  Rey Follow-up | 0.23 (1.23) | 0.22 (0.89) | -0.09 (1.00) | 0.44 (1.14)

31. Secondary Outcome: Miami Instrumental Activities of Daily Living Task Post Training
Description: Score on Miami Instrumental Activities of Daily Living task, at baseline and immediately after 4 weeks of training, based on number of correct tasks/time completed. Higher scores represent more tasks completed per minute, and therefore better performance. Scores have a minimum of 0, and no set maximum.
Time Frame: Baseline, Immediately after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tasks completed per minute
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 49 | 47 | 50 | 56
Tasks completed per minute
  ATM Task Baseline | 3.17 (1.32) | 2.78 (1.03) | 2.67 (1.20) | 2.81 (1.13)
  ATM Task Post Training | 3.19 (1.07) | 3.23 (1.01) | 2.98 (1.07) | 2.97 (1.10)
  Prescription Task Baseline | 4.31 (4.54) | 3.67 (1.44) | 3.54 (1.32) | 3.40 (1.50)
  Prescription Task Post Training | 4.75 (2.49) | 4.91 (5.43) | 4.20 (1.58) | 4.14 (3.15)

32. Secondary Outcome: Miami Instrumental Activities of Daily Living Task at One Year
Description: Score on Miami Instrumental Activities of Daily Living task, at baseline and one year after 4 weeks of training, based on number of correct tasks/time completed. Higher scores represent more tasks completed per minute, and therefore better performance. Scores have a minimum of 0, and no set maximum.
Time Frame: Baseline, One-year after 4-week intervention training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tasks completed per minute
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
Number analyzed (Participants) | 45 | 37 | 40 | 47
Tasks completed per minute
  ATM Task Baseline | 3.18 (1.31) | 3.03 (0.94) | 2.78 (1.19) | 2.79 (1.13)
  ATM Task Follow-up | 3.09 (1.11) | 3.26 (1.14) | 3.12 (1.26) | 2.85 (1.04)
  Prescription Task Baseline | 4.40 (4.72) | 3.72 (1.39) | 3.65 (1.30) | 3.40 (1.47)
  Prescription Task Follow-up | 4.22 (2.31) | 3.98 (1.09) | 4.08 (2.13) | 4.26 (2.04)

ADVERSE EVENTS:
Time Frame: From enrollment to the end of the follow-up assessment (approx. 1 year)
Arm/Group | BrainHQ | Rise of Nations | IADL Training | Active Control
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/59 | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/59 | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 0/57 | 0/59 | 0/56 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03141281/Prot_002.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT03141281/SAP_003.pdf
  • Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03141281/ICF_000.pdf